CLINICAL TRIAL: NCT03130933
Title: Does a Single Dose of Systemic Antibiotics Prevent Postoperative Inflammatory Complications After Lower Third Molar Surgery? A Randomized Controlled Trial
Brief Title: Complications After Lower Third Molar Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Ana Kotarac Knežević, Principal investigator, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCHOOL OF DENTAL MEDICINE
Record Dates: First submitted 2017-04-17; First posted 2017-04-27 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Postoperative Complications; Third Molar
Keywords: third molar; oral surgical procedures; antibiotic prophylaxis; placebo effect
MeSH Terms: conditions — Postoperative Complications | interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: A RANDOMIZED CONTROLLED TRIAL
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There was 400 participiants, patients and the same oral surgeon
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The first tested subgroup (Active Comparator): The tested subgroup from the main group without prior inflammation received a prophylactic single dose of 4 x Amoxicillin 500 Mg one hour prior the lower third molar surgery.
  Interventions: Procedure: Lower third molar surgery; Drug: Amoxicillin 500 Mg
- The first control subgroup (Placebo Comparator): The control subgroup from the main group without prior inflammation received a placebo one hour prior the lower third molar surgery .
  Interventions: Procedure: Lower third molar surgery; Other: Placebo
- The second tested subgroup (Active Comparator): The tested subgroup from the main group with prior inflammation received a prophylactic single dose of 4 x Amoxicillin 500 Mg one hour prior the lower third molar surgery .
  Interventions: Procedure: Lower third molar surgery; Drug: Amoxicillin 500 Mg
- The second control subgroup (Placebo Comparator): The control subgroup from the main group with prior inflammation received a placebo one hour prior the lower third molar surgery .
  Interventions: Procedure: Lower third molar surgery; Other: Placebo

INTERVENTIONS:
Procedure: Lower third molar surgery — All surgical procedures were performed under local anaesthesia (alveolar nerve block) with 2% lidocaine chloride. The full-thickness mucoperiosteal flap was raised using buccal approach, adequate osteotomy was done using micromotor handpiece and bur, and third molar removal was finished using elevating instruments in the appropriate direction. Removal of bone dust, granulation tissue and broken tooth fragments were done in order to wound toileting. Gentle, sterile saline irrigation was done on the end.
  Primary closure of the surgical area was done using 3-0 silk sutures.
Drug: Amoxicillin 500 Mg — The tested subgroups received a prophylactic single dose of 4 x 500 Mg Amoxicillin one hour prior the lower third molar surgery.
  Other Names: prophylaxis
  Arms: The first tested subgroup; The second tested subgroup
Other: Placebo — The control subgroups received a prophylactic single dose of placebo one hour prior the lower third molar surgery.
  Arms: The first control subgroup; The second control subgroup

SUMMARY:
Objectives: The objective of the study was to evaluate the effectiveness of a prophylactic single preoperative dose of amoxicillin in decreasing complications after lower third molar surgery.

Materials and methods: The sample consisted of 400 patients randomly divided in two groups consisting of 200 patients per each group. The patients underwent third molar surgery at the Department of Oral Surgery, Clinical Hospital Dubrava, Croatia, in the period between April 2010. and November 2016. Unlike the patients from the second group, the first group of patients had never been diagnosed inflammation prior the surgical procedure. The main tested groups were further divided in two subgroups (control and tested): the tested subgroup (100 patients) received a prophylactic single dose of 2 g amoxicillin an hour prior the procedure, while the second control subgroup (100 patients) received a placebo. Complications, including swelling, alveolar osteitis (AO), infection at the surgical site (SSI), limited mouth opening, pain, bleeding, and increased body temperature, were evaluated postoperatively. Evaluation was done on the first postoperative day and 7 days after surgery.

DETAILED DESCRIPTION:
Study design and sample description This prospective study was performed at the Department of Oral Surgery of Clinical Hospital Dubrava, Zagreb, Croatia, in the period from April 2010. through November 2016. All patients voluntarily agreed and written consent to participate in the study was obtained from each participant. The study was approved by Ethics Committee of the School of Dental Medicine, Zagreb, Croatia (81-2009). The identity of the subjects was protected in all phases of the study.

The exclusion criteria in this study were systematic diseases, with developing local infections, current smokers, pregnant women, lactating females, patients using oral contraceptive drugs and those under any antibiotic coverage.

The sample consisted of systematically healthy subjects between 18 to 40 years (both gender) and having semi-impacted lower third molars indicated for surgical removal randomly divided into two main groups of patients. Unlike the patients from the second group, the first group of patients had never been diagnosed inflammation prior the surgical procedure. The main tested groups were further divided in two subgroups (control and tested): the tested subgroup (100 patients) received a prophylactic single dose of 2 g amoxicillin an hour prior the procedure, while the second control subgroup (100 patients) received a placebo. The selection of third molars for control and study subgroup was made according to Pederson difficulty index (9). According to this index (Table 1), the patients are classified into 3 groups: easy, moderate and difficult. The patients from this study who were classified into a difficult group were excluded from the study due to a longer and complicated surgical procedure with an expected prolonged recovery period and possible postoperative complications.

The patients were recalled for follow-up on post-operative days one and seven. In all tested groups data had been obtained by using identical questionnaire. The following symptoms were assessed: pain, swelling, wound healing (AO, SSI), maximum inter-incisal opening of mouth, increased body temperature and hemorrhage. A postoperative follow-up was done always by the single experienced therapist. Patients evaluated their postoperative pain with grades from 0-10 using according to visual analogue scale (VAS) where the end points were marked as "no pain" (0) and "unbearable pain" (10). Surgeon evaluated the type of post-extraction alveolus healing as following normal healing, acute inflammation followed by infected alveolus and dry socket. The surgeon who assessed wound swelling did not know to which group the patient was allocated. The method of assessing the swelling was described in our previous study (10). The post-operative swelling was assessed on postoperative days 1 and 7, using four-point scale as 0=no swelling, 1=mild swelling, 2=moderate swelling, 3=severe swelling.

The maximum inter-incisal opening of the mouth was calculated from the mesioincisal angle of the ipsilateral mandibular central incisor to the mesioincisal angle of the ipsilateral mandibular central incisor using digital calliper (Caliper-Digital; Salvin Dental Specialties, Inc, Charlotte, NC).

Increased body temperature was measured by patient at home during postoperative period of seven days. Body temperature within 36.0ºC and 37.5ºC was evaluated as normal. The body temperature under 37.5 ºC was evaluated as increased. All temperatures were measured at the same time of the day, between 9:00 and 11:00 a.m.

Hemorrhage was observed by patient during next seven days after the surgical procedure. It was classified as absent or present through following days. Present hemorrhage was classified as light or intense.

The outcome variable was the presence or absence of an inflammatory complication after third molar surgery (SSI or AO). A diagnosis of SSI was identified by purulent discharge from the surgical site at any point postoperatively, fever, lymphadenopathy, or pain and edema warranting surgical intervention and/or systematic antibiotics. Alveolar osteitis was diagnosed in cases of an empty alveolar socket, increasing pain lasting more than 2 days after surgery, and exposed alveolar bone tissue.

ELIGIBILITY:
Inclusion Criteria:

* systematically healthy subjects between 18 to 40 years (both gender) and having semi-impacted lower third molars indicated for surgical removal

Exclusion Criteria:

* The exclusion criteria in this study were systematic diseases, with developing local infections, current smokers, pregnant women, lactating females, patients using oral contraceptive drugs and those under any antibiotic coverage.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pain | 1 day and 7 days after surgery
  Patients evaluated their postoperative pain with grades from 0-10 using according to visual analogue scale (VAS) where the end points were marked as "no pain" (0) and "unbearable pain"(10).

SECONDARY OUTCOMES:
Swelling | 1 day and 7 days after surgery
  The post-operative swelling was assessed on postoperative days 1 and 7, using four-point scale as 0=no swelling, 1=mild swelling, 2=moderate swelling, 3=severe swelling.
Wound healing ( AO, SSI ) | 1 day and 7 days after surgery
  Surgeon evaluated the type of post-extraction alveolus healing as following normal healing, acute inflammation followed by infected alveolus and dry socket.
Maximum inter-incisal opening of mouth | 1 day and 7 days after surgery
  The maximum inter-incisal opening of the mouth was calculated from the mesioincisal angle of the ipsilateral mandibular central incisor to the mesioincisal angle of the ipsilateral mandibular central incisor using digital calliper (Caliper-Digital; Salvin Dental Specialties, Inc, Charlotte, NC).
Increased body temperature | through 7 days
  Increased body temperature was measured by patient at home during postoperative period of seven days. Body temperature within 36.0ºC and 37.5ºC was evaluated as normal. The body temperature under 37.5 ºC was evaluated as increased. All temperatures were measured at the same time of the day, between 9:00 and 11:00 a.m.
Hemorrhage | through 7 days
  Hemorrhage was observed by patient during next seven days after the surgical procedure. It was classified as absent or present through following days. Present hemorrhage was classified as light or intense.

CONTACTS AND LOCATIONS:
Overall Officials: Marko Granić, DMD,PhD, Study Chair — Second author; Tihomir Kuna, DMD, PhD, Study Chair — Third author; Dinko Knežević, DMD, Study Chair — fourth author; Nino Grgić, DMD, Study Chair — fifth author
Locations (1):
- School of dental medicine, University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bahl R, Sandhu S, Singh K, Sahai N, Gupta M. Odontogenic infections: Microbiology and management. Contemp Clin Dent. 2014 Jul;5(3):307-11. doi: 10.4103/0976-237X.137921. PMID 25191064
- [Result] Chuang SK, Perrott DH, Susarla SM, Dodson TB. Risk factors for inflammatory complications following third molar surgery in adults. J Oral Maxillofac Surg. 2008 Nov;66(11):2213-8. doi: 10.1016/j.joms.2008.06.067. PMID 18940482
- [Result] Baqain ZH, Karaky AA, Sawair F, Khraisat A, Duaibis R, Rajab LD. Frequency estimates and risk factors for postoperative morbidity after third molar removal: a prospective cohort study. J Oral Maxillofac Surg. 2008 Nov;66(11):2276-83. doi: 10.1016/j.joms.2008.06.047. PMID 18940492
- [Result] Chuang SK, Perrott DH, Susarla SM, Dodson TB. Age as a risk factor for third molar surgery complications. J Oral Maxillofac Surg. 2007 Sep;65(9):1685-92. doi: 10.1016/j.joms.2007.04.019. PMID 17719384
- [Result] Arteagoitia MI, Barbier L, Santamaria J, Santamaria G, Ramos E. Efficacy of amoxicillin and amoxicillin/clavulanic acid in the prevention of infection and dry socket after third molar extraction. A systematic review and meta-analysis. Med Oral Patol Oral Cir Bucal. 2016 Jul 1;21(4):e494-504. doi: 10.4317/medoral.21139. PMID 26946211
- [Result] Seymour RA, Walton JG. Pain control after third molar surgery. Int J Oral Surg. 1984 Dec;13(6):457-85. doi: 10.1016/s0300-9785(84)80017-4. PMID 6150903
- [Result] Batinjan G, Zore Z, Celebic A, Papic M, Gabric Panduric D, Filipovic Zore I. Thermographic monitoring of wound healing and oral health-related quality of life in patients treated with laser (aPDT) after impacted mandibular third molar removal. Int J Oral Maxillofac Surg. 2014 Dec;43(12):1503-8. doi: 10.1016/j.ijom.2014.09.003. Epub 2014 Sep 29. PMID 25277807
- [Result] Dodson TB. HIV status and the risk of post-extraction complications. J Dent Res. 1997 Oct;76(10):1644-52. doi: 10.1177/00220345970760100501. PMID 9326896
- [Result] Dodson TB. Predictors of postextraction complications in HIV-positive patients. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1997 Nov;84(5):474-9. doi: 10.1016/s1079-2104(97)90260-2. PMID 9394376
- [Result] Halpern LR, Dodson TB. Does prophylactic administration of systemic antibiotics prevent postoperative inflammatory complications after third molar surgery? J Oral Maxillofac Surg. 2007 Feb;65(2):177-85. doi: 10.1016/j.joms.2006.10.016. PMID 17236918
- [Result] Falconer DT, Roberts EE. Report of an audit into third molar exodontia. Br J Oral Maxillofac Surg. 1992 Jun;30(3):183-5. doi: 10.1016/0266-4356(92)90154-b. PMID 1622965
- [Result] Crincoli V, Di Comite M, Di Bisceglie MB, Petruzzi M, Fatone L, De Biase C, Tecco S, Festa F. Which route of antibiotic administration should be used for third molar surgery? A split-mouth study to compare intramuscular and oral intake. Clin Ter. 2014;165(1):e12-6. doi: 10.7471/CT.2014.1665. PMID 24589954
- [Result] Lockhart PB, Brennan MT, Kent ML, Norton HJ, Weinrib DA. Impact of amoxicillin prophylaxis on the incidence, nature, and duration of bacteremia in children after intubation and dental procedures. Circulation. 2004 Jun 15;109(23):2878-84. doi: 10.1161/01.CIR.0000129303.90488.29. Epub 2004 Jun 1. PMID 15173031
- [Result] Hall G, Nord CE, Heimdahl A. Elimination of bacteraemia after dental extraction: comparison of erythromycin and clindamycin for prophylaxis of infective endocarditis. J Antimicrob Chemother. 1996 Apr;37(4):783-95. doi: 10.1093/jac/37.4.783. PMID 8722544
- [Result] Yoshii T, Hamamoto Y, Muraoka S, Furudoi S, Komori T. Differences in postoperative morbidity rates, including infection and dry socket, and differences in the healing process after mandibular third molar surgery in patients receiving 1-day or 3-day prophylaxis with lenampicillin. J Infect Chemother. 2002 Mar;8(1):87-93. doi: 10.1007/s101560200012. PMID 11957126
- [Result] Monaco G, Tavernese L, Agostini R, Marchetti C. Evaluation of antibiotic prophylaxis in reducing postoperative infection after mandibular third molar extraction in young patients. J Oral Maxillofac Surg. 2009 Jul;67(7):1467-72. doi: 10.1016/j.joms.2008.12.066. PMID 19531419
- [Result] Esposito S, Novelli A, de Lalla F. [Antibiotic prophylaxis in surgery: news and controversies]. Infez Med. 2002 Sep;10(3):131-44. Italian. PMID 12704263
- [Result] Lee JY, Do HS, Lim JH, Jang HS, Rim JS, Kwon JJ, Lee ES. Correlation of antibiotic prophylaxis and difficulty of extraction with postoperative inflammatory complications in the lower third molar surgery. Br J Oral Maxillofac Surg. 2014 Jan;52(1):54-7. doi: 10.1016/j.bjoms.2013.08.010. Epub 2013 Sep 9. PMID 24029441
- [Result] Alanis A, Weinstein AJ. Adverse reactions associated with the use of oral penicillins and cephalosporins. Med Clin North Am. 1983 Jan;67(1):113-29. doi: 10.1016/s0025-7125(16)31227-5. No abstract available. PMID 6219257
- [Result] Hawkey PM, Patel BC, Trees AJ. UK antimicrobial resistance strategy must be set in a wider context. BMJ. 2013 May 15;346:f2999. doi: 10.1136/bmj.f2999. No abstract available. PMID 23678076
- [Result] Marcussen KB, Laulund AS, Jorgensen HL, Pinholt EM. A Systematic Review on Effect of Single-Dose Preoperative Antibiotics at Surgical Osteotomy Extraction of Lower Third Molars. J Oral Maxillofac Surg. 2016 Apr;74(4):693-703. doi: 10.1016/j.joms.2015.11.017. Epub 2015 Nov 23. PMID 26706491
- [Result] Conrad SM, Blakey GH, Shugars DA, Marciani RD, Phillips C, White RP Jr. Patients' perception of recovery after third molar surgery. J Oral Maxillofac Surg. 1999 Nov;57(11):1288-94; discussion 1295-6. doi: 10.1016/s0278-2391(99)90861-3. PMID 10555792
- [Result] Phillips C, White RP Jr, Shugars DA, Zhou X. Risk factors associated with prolonged recovery and delayed healing after third molar surgery. J Oral Maxillofac Surg. 2003 Dec;61(12):1436-48. doi: 10.1016/j.joms.2003.08.003. PMID 14663809
- [Result] Phillips C, Gelesko S, Proffit WR, White RP Jr. Recovery after third-molar surgery: the effects of age and sex. Am J Orthod Dentofacial Orthop. 2010 Dec;138(6):700.e1-8; discussion 700-1. doi: 10.1016/j.ajodo.2010.06.013. PMID 21130316
- [Result] Blondeau F, Daniel NG. Extraction of impacted mandibular third molars: postoperative complications and their risk factors. J Can Dent Assoc. 2007 May;73(4):325. PMID 17484797
- [Result] Waite PD, Cherala S. Surgical outcomes for suture-less surgery in 366 impacted third molar patients. J Oral Maxillofac Surg. 2006 Apr;64(4):669-73. doi: 10.1016/j.joms.2005.12.014. PMID 16546647
- [Result] Ren YF, Malmstrom HS. Effectiveness of antibiotic prophylaxis in third molar surgery: a meta-analysis of randomized controlled clinical trials. J Oral Maxillofac Surg. 2007 Oct;65(10):1909-21. doi: 10.1016/j.joms.2007.03.004. PMID 17884515
- [Result] Lodi G, Figini L, Sardella A, Carrassi A, Del Fabbro M, Furness S. Antibiotics to prevent complications following tooth extractions. Cochrane Database Syst Rev. 2012 Nov 14;11:CD003811. doi: 10.1002/14651858.CD003811.pub2. PMID 23152221
- [Result] Bortoluzzi MC, Capella DL, Barbieri T, Pagliarini M, Cavalieri T, Manfro R. A single dose of amoxicillin and dexamethasone for prevention of postoperative complications in third molar surgery: a randomized, double-blind, placebo controlled clinical trial. J Clin Med Res. 2013 Feb;5(1):26-33. doi: 10.4021/jocmr1160w. Epub 2013 Jan 11. PMID 23390473
- [Result] Pasupathy S, Alexander M. Antibiotic prophylaxis in third molar surgery. J Craniofac Surg. 2011 Mar;22(2):551-3. doi: 10.1097/SCS.0b013e31820745c7. PMID 21403575
- [Result] Isiordia-Espinoza MA, Aragon-Martinez OH, Martinez-Morales JF, Zapata-Morales JR. Risk of wound infection and safety profile of amoxicillin in healthy patients which required third molar surgery: a systematic review and meta-analysis. Br J Oral Maxillofac Surg. 2015 Nov;53(9):796-804. doi: 10.1016/j.bjoms.2015.06.013. Epub 2015 Aug 25. PMID 26316017
- [Result] Lopez-Cedrun JL, Pijoan JI, Fernandez S, Santamaria J, Hernandez G. Efficacy of amoxicillin treatment in preventing postoperative complications in patients undergoing third molar surgery: a prospective, randomized, double-blind controlled study. J Oral Maxillofac Surg. 2011 Jun;69(6):e5-14. doi: 10.1016/j.joms.2011.01.019. Epub 2011 Apr 5. PMID 21470751
- [Result] Ong CK, Seymour RA. Pathogenesis of postoperative oral surgical pain. Anesth Prog. 2003 Winter;50(1):5-17. PMID 12722900
- See also: Conaty S, Hoang H, Kirshen D, Kwong C, Schroeder E, Stromme A: Pre and post-operative antibiotic prophylaxis in the prevention of complications following third molars surgery — http://docplayer.net/29390208-Pre-and-post-operative-antibiotic-prophylaxis-in-the-prevention-of-complications-following-third-molar-surgery.html#show_full_text